CLINICAL TRIAL: NCT02362334
Title: Precision of Optical Biometry and Intraocular Lens Power Calculation Using Dual Schiempflug Analyzer
Brief Title: IOL Power Calculation Using Dual Schiempflug Analyzer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChuncheonSHH
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-10

CONDITIONS: Cataract
Keywords: dual Sheimpflug analyzer; intraocular lens power; optical low-coherence reflectometry
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the various ocular parameters which are necessary for ocular biometry and the calculated IOL powers using both dual Schiempflug analyzer and optical low-coherence refelctometry.

DETAILED DESCRIPTION:
The measured keratometry, axial length, anterior chamber depth, lens thickness, white-to-white corneal diameter, and calculated IOL powers using various formulas including Hoffer Q, Holladay I, SRK II and SRK T measured by dual Schiempflug analyzer and optical low-coherence refelctometry will be compared.

ELIGIBILITY:
Inclusion Criteria:

* axial length between 21.0 and 27.0 mm
* older than 20 years old

Exclusion Criteria:

* other ophthalmic diseases such as severe dry eye, glaucoma, and age-related macular degeneration
* previous ophthalmic surgery including cataract surgery, and refractive surgery
* very dense media which cannot be measured by the optical biometries
* severe zonulysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 140 eyes of patients who scheduled for cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Ocular parameters | Single point
  Parameters measured using two devices were compared at a single point
Calculated IOL powers | Single point
  Calculated IOL powers using two devices were compared at a single point

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Eun Han, MD, Study Chair — Clinical associate professor
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, South Korea